CLINICAL TRIAL: NCT05908175
Title: FES-assisted Gait Training Intervention to Improve Gait in Individuals with an Incomplete Spinal Cord Injury - a Pilot Study
Brief Title: FES-assisted Gait Intervention in People with Spinal Cord Injury - Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stichting Reade (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W23.009; NL82880.015.22 (Other: CCMO)
Record Dates: First submitted 2023-05-08; First posted 2023-06-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Other): FES-assisted gait training intervention group
  Interventions: Other: FES-assisted gait training

INTERVENTIONS:
Other: FES-assisted gait training — The participants will walk with functional electrical stimulation (and possible body weight support) on a treadmill for 10 weeks, twice a week for 30 minutes.

SUMMARY:
A spinal cord injury (SCI) disrupts the communication within the nervous system, leading to limitations in sensorimotor activities such as walking. Regular use of functional electrical stimulation (FES) can result in recovery of voluntary muscle control and muscle strength. Locomotor training with FES may be a promising method to improve gait function. The primary objective of this pilot study is to assess the feasibility and safety of an FES-assisted gait training intervention. Secondary objectives are to assess the effects of an FES-assisted gait training intervention on gait function.

DETAILED DESCRIPTION:
A spinal cord injury (SCI) disrupts the communication within the nervous system, leading to limitations in sensorimotor activities, such as walking. These limitations are associated with muscle weakness, a disturbance of the reflex activity, and the inability or difficulty to recruit muscles below the lesion. Regular use of functional electrical stimulation (FES) can result in recovery of voluntary muscle control and muscle strength. Studies that investigated the effect of locomotor training on a treadmill with functional electrical stimulation and/or body weight support (BWS) show improved function of the lower limbs. FES-assisted gait therapy may be a promising method for improving gait function in individuals with an incomplete SCI. Therefore, this study will investigate if an FES-assisted gait (with BWS) is feasible and safe. This study will also investigfate if an FES-assisted gait can improve gait function in people with an incomplete SCI.

Primary objective of this pilot study is to assess the feasibility and safety of an FES-assisted gait training intervention. The secondary objectives are to assess the effects of an FES-assisted gait training intervention on gait function.

ELIGIBILITY:
Inclusion Criteria:

* Have a non-progressive incomplete SCI.
* Have limited motor abilities in the lower extremities.
* Be able to walk on a treadmill for 30 minutes (with body weight support).
* Be able to perform the 10 meter walk test overground with assistive devices and/or support form the researcher/physician.
* Have a stable medical condition.
* Have had the SCI for at least a year.
* Be at least 18 years of age.

Exclusion Criteria:

* Cardiac arrhythmias or cardiac disease;
* Flaccid paralysis.
* Musculoskeletal dysfunction, uncured fractures, contractures, pressure injuries, or infections that could impede the intended training;
* A history of severe autonomic dysreflexia assessed with the 'Autonomic standards assessment';
* Neurostimulator, pacemaker, or other device that prevents the safe use of electrical stimulation present in the body;
* Very high sensitivity to electrical stimulation, i.e., sensitivity threshold is reached before motor responses are observed in all target muscles;
* Insufficient mastery of the Dutch language (speaking and reading);
* Severe cognitive or communicative disorders;
* Being or becoming pregnant during the study period;
* Severe psychiatric illness or disorders (at the discretion of the treating rehabilitation physician);
* Involved in another intervention study which may have an effect on the outcome measures of the present study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention | Assessed during week 11 during the post-intervention measurement.
  Self-administered questionnaires about the training sessions, preceived effect, applicability of FES and the experience with walking with FES.
Incidence of (Serious) Adverse Events [Safety of the Intervention] | Assessed during week 1 to 10 for each FES-assisted gait training session (2x week) and in week 0, week 11 and week 21 (during the pre-, post- and follow-up measurements)
  The total number of (serious) adverse events

SECONDARY OUTCOMES:
Change in average and maximum treadmill walking speed | Assessed during each FES-assisted gait training session (from week 1 until week 10, 2x a week)
  Average and maximum walking speed (m/s) recorded by the treadmill during each training session
Change in distance | Assessed during each FES-assisted gait training session (from week 1 until week 10, 2x a week)
  Distance (in meters) recorded by the treadmill during each training session.
Change in average overground walking speed | Assessed before and after the 10-weeks FES-assisted gait training intervention (during week 0 and week 11)
  Walking speed (m/s) measured by 10 meter walk test
Change in muscle activity | Assessed before and after the 10-weeks FES-assisted gait training intervention (during week 0 and week 11)
  Surface EMG measurement during 10 meter walk test. Time of muscle activation and duration of muscle activity of the m. rectus femoris, m. vastus lateralis, m. semitendinosus, m. tibialis anterior, m. gastrocnemius medialis, m. soleus and m. peroneus longus
Change in step length | Assessed before and after the 10-weeks FES-assisted gait training intervention (during week 0 and week 11)
  Step length left and right (cm) measured during 10 meter walk test with the interactive walkway (kinect)
Change in step width | Assessed before and after the 10-weeks FES-assisted gait training intervention (during week 0 and week 11)
  Step width (cm) measured during 10 meter walk test with interactive walkway (kinect)
Change in cadence | Assessed before and after the 10-weeks FES-assisted gait training intervention (during week 0 and week 11)
  Cadence (steps/min) measured during 10 meter walk test with interactive walkway (kinect)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Janssen, Prof. Dr., Principal Investigator — Stichting Reade
Locations (1):
- Stichting Reade, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No